CLINICAL TRIAL: NCT00002108
Title: 3TC (Lamivudine; GR109714X) Open-Label Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Glaxo Wellcome (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: None | Purpose: Treatment
Other Study IDs: 129D; NUCA 3004
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1995-11

CONDITIONS: HIV Infections
Keywords: Drug Therapy, Combination; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Antiviral Agents; Zidovudine
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Lamivudine; Zidovudine

INTERVENTIONS:
Drug: Lamivudine
Drug: Zidovudine

SUMMARY:
To make lamivudine (3TC) available to patients with progressive, symptomatic HIV disease who cannot participate in a controlled clinical trial and who are refractory or unable to tolerate other therapies. To collect data pertaining to the safety of 3TC at two dose levels. To evaluate the effect of 3TC on markers of hepatitis B in co-infected patients at five to ten selected sites.

DETAILED DESCRIPTION:
Patients 12 years and older are randomized to receive one of two doses of 3TC for a duration determined by the patient's physician or until termination of the program. Patients < 12 years receive a lower dose of 3TC. Patients are followed monthly. For selected sites only, serum samples are collected every 3 months from patients identified as HBsAg positive.

PER 02/28/95 AMENDMENT: Patients enrolled prior to 3/1/95 may remain on their assigned monotherapy dose or change to combination therapy with 3TC and zidovudine.

ELIGIBILITY:
Patients must:

* Have progressive, symptomatic HIV disease.
* Have a mean CD4 count <= 99 cells/mm3 for adults and <= 300 cells/mm3 for children (original design was CD4 count <= 300 cells/mm3 for both adults and children).
* Be unable to participate in a controlled trial.
* Be refractory to or unable to tolerate other therapies.
* Be able to attend clinic on a monthly schedule.
* Have consent of parent or guardian if under the age of consent.

NOTE:

* If a pregnant or breast-feeding woman requests enrollment, her physician should contact Glaxo staff directly to discuss the case.

Practice of unsafe sex.

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Kern - McNeill International, Morristown, New Jersey, United States

REFERENCES:
- [Background] Pluda J, Cooley T, Montaner J, McCaffrey R, Wainberg M, Yarchoan R. Phase I/II study of 3TC (GR109714X) in adults with ARC or AIDS. Int Conf AIDS. 1993 Jun 6-11;9(1):69 (abstract no WS-B26-2)